CLINICAL TRIAL: NCT01124955
Title: Acupuncture for Acute Nonspecific Low Back Pain: a Randomized, Controlled, Double-blind, Placebo Trial
Brief Title: Acupuncture Using Yamamoto's Method for the Treatment of Acute Nonspecific Low Back Pain
Acronym: ANLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Tatiana Molinas Hasegawa, Federal University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDAAAAU
Record Dates: First submitted 2010-05-13; First posted 2010-05-18 (Estimated); Results first posted 2011-06-13 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2009-11

CONDITIONS: Low Back Pain
Keywords: treatment; acupuncture; spine
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Active Comparator): Patients receive 5 sessions of real acupuncture. The technique of acupuncture used in this study is Yamamoto New Scalp Acupuncture called YNSA.
  Interventions: Other: Acupuncture
- Non-penetrating acupuncture (Placebo Comparator): The placebo group (PG) are submitted to five non-penetrating acupuncture sessions using YNSA.
  Interventions: Other: Non-penetrating acupuncture

INTERVENTIONS:
Other: Acupuncture — The intervention group (IG) are submitted to five acupuncture sessions using Yamamoto New Scalp Acupuncture(YNSA)
  Other Names: Real acupuncture
  Arms: Intervention Group
Other: Non-penetrating acupuncture — The placebo group (PG) are submitted to five non-penetrating acupuncture sessions using YNSA.
  Other Names: Placebo acupuncture
  Arms: Non-penetrating acupuncture

SUMMARY:
The aim of the present study is to assess the effectiveness of acupuncture using Yamamoto's method for the treatment of ANLBP using the following outcomes:pain,functional capacity,quality of life and number of 50 mg sodium diclofenac pills taken per day.

DETAILED DESCRIPTION:
A randomized, controlled, double-blind, prospective trial is being conducted involving 80 patients with low-back pain defined as pain and discomfort localised bellow the costal margin and above the inferior gluteal folds, for a period of less than 30 days and unrelated to any specific etiological factors. Patients are being recruited from the university hospital of the Federal University of Sao Paul (UNIFESP)and exams were carried out by a rheumatologist. The patients are randomly assigned to either intervention group (IG) and are submitted to five acupuncture sessions or placebo group (PG) and are submitted to five non-penetrating acupuncture sessions. Both groups are recommended to take 50 mg of sodium diclofenac every eight hours for lumbar pain, if needed and record the number of pills on a standardized form.

The patients are instructed not to use other medications or therapies for low-back pain during the study.The IG are submitted to acupuncture by a physician acupuncturist with eight years experience in the technique. Five acupuncture session are performed at baseline, D3, D7, D14 and D21. Specific needles for scalp acupuncture and tubes that guide these needles, called mandrels are unpacked in front of the patient. The stainless steel needles: 0.20 x 13 mm, sterilized and disposable.Sessions last 20 minutes. The patient remain seated, using a hat with a central orifice exposing the area to receive the needles. The hat has a wide brim to keep the patient blinded for the procedures. The needle penetrates the skin at an approximately 15º angle and a depth of 0.3 to 0.5 cm. The PG are submitted to five placebo acupuncture session performed by the same acupuncturist with same material and hat, but penetration did not occur and only the mandrel came into contact with the skin. All patients are blind to which procedure they are receiving. The basic points D, H and I and kidney, bladder and liver points of Yamamoto's method are used as standard treatment to ANLBP for the both groups.

Evaluations: The IG and PG are evaluated six times between baseline and Day 28 immediately before and after each acupuncture session. Outcome measures are recorded by a single assessor blinded to group allocation.

D0: baseline; D3: three days after baseline; D7: seven days after baseline; D14: fourteen days after baseline; D21: twenty-one days after baseline and D28: twenty-eight days after baseline.

Losses: Participants absent from more than three acupuncture sessions and evaluations are considered losses.

Placebo credibility: At the end of the study, participants are asked about which group they believed they belonged.

Sample size: To achieve an improvement in VAS pain of 2.0 point, with a significance of 0.05, and a power of 0.90, a minimum of 40 patients per group is necessary as a previous compensation for the possible 20% loss at follow-up.

Statistics: An intention-to-treat analysis are performed, using the last-observation-carried-forward method. A level of significance of p < 0.05 (2-tailed tests) are accepted for the trial. For normally distributed data, the variables are analysed using repeated-measures analysis of variance (ANOVA). The analysis are performed between groups (acupuncture versus non-penetrating acupuncture; between subjects factors) and over the time (baseline, 3, 7, 14, 21 and 28 days; within subjects factors). Categorical data measured over time are analysed using repeated-measures analyses of variance (ANOVA) for categorical data. A 95% confidence interval (95% CI) are used. The Student's t-test are used to compare numerical variables with normal distribution at one time and the chi-square test or Fisher's exact test are used to determine differences in rates of improvement between the two groups. The Kappa index are used to determine agreement on the LIKERT assessment between patient and assessor. All tests are performed using SPSS version 15.0 and MINITAB 14.0

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18 to 65 years
* Seeking medical assistance for nonspecific low-back pain
* Score of 4 to 8 cm on the pain scale (0 to 10 cm)
* Agreed to participate and signed term of informed consent

Exclusion Criteria:

* Patients with a diagnostic investigation of secondary causes as spondyloarthropathy, infection, tumor or fracture
* Sciatica lumbar pain
* Previous surgery on spinal column
* Litigation
* Having changed physical activity or underwent acupuncture or physical therapy in previous three months,
* Having previously undergone scalp acupuncture
* Pregnancy
* Contraindication for anti-inflammatory agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, MD,PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Tatiana Hasegawa, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Inoue M, Hojo T, Nakajima M, Kitakoji H, Itoi M. Comparison of the effectiveness of acupuncture treatment and local anaesthetic injection for low back pain: a randomised controlled clinical trial. Acupunct Med. 2009 Dec;27(4):174-7. doi: 10.1136/aim.2009.001164. PMID 19942724
- [Derived] Hasegawa TM, Baptista AS, de Souza MC, Yoshizumi AM, Natour J. Acupuncture for acute non-specific low back pain: a randomised, controlled, double-blind, placebo trial. Acupunct Med. 2014 Apr;32(2):109-15. doi: 10.1136/acupmed-2013-010333. Epub 2013 Dec 6. PMID 24316509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 patients were recruited from the university hospital of the Federal University of São Paul (UNIFESP), from November 2009 to June 2010.
Pre-assignment Details: 80 patients were randomized during the study.
Groups:
- Acupuncture: The technique of acupuncture used in this study is Yamamoto New Scalp Acupuncture called YNSA.
- Placebo Group: Patients were submitted to five non-penetrating acupuncture sessions in the placebo group (PG).
Period: Overall Study
Arm/Group | Acupuncture | Placebo Group
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Placebo Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  Between 18 and 65 years | 40 | 40 | 80
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (9.8) | 43.9 (10.9) | 45.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  Brazil | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessed on a 10-point Numeric Pain Scale
Description: The primary outcome is a visual analog pain scale (VAS), graded in centimeters from 0 to 10 (0=no pain; 10=worst imaginable pain), measured before (VAS 1) and after (VAS 2) the acupuncture session.
Time Frame: days 0, 3, 7, 14, 21 and 28
Population: Intention to treat analysis (ITT)
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: cm
Arm/Group | Acupuncture | Placebo Group
Number analyzed (Participants) | 40 | 40
Number analyzed (cm) | 40 | 40
cm
  Day 0 | 6.55 (1.4) | 6.68 (1.44)
  Day 3 | 4.63 (2.23) | 5.13 (2.21)
  Day 7 | 3.83 (2.61) | 4.4 (2.09)
  Day 14 | 2.8 (2.27) | 3.95 (2.19)
  Day 21 | 2.49 (2.4) | 4.18 (2.52)
  Day 28 | 1.98 (2.12) | 3.38 (2.26)

2. Secondary Outcome: Roland-Morris Disability Questionnaire (RM)
Description: Secondary outcomes includes the Roland-Morris Disability Questionnaire (RM) for the assessment of functional capacity, with 24 items on low-back pain: higher scores denote poorer functional capacity.
  0: better functional capacity 24: poorer functional capacity Range of score: the highest is 24 (poorer functional capacity) and lowest scores is 0 (better functional capacity).
Time Frame: days 0, 3, 7, 14, 21 and 28
Population: Intention to treat analysis (ITT)
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Acupuncture | Placebo Group
Number analyzed (Participants) | 40 | 40
Number analyzed (scores on a scale) | 40 | 40
scores on a scale
  Day 0 | 14.9 (4.0) | 14.6 (4.8)
  Day 3 | 10.3 (5.4) | 12.4 (4.5)
  Day 7 | 8.1 (5.5) | 10.2 (5.3)
  Day14 | 5.3 (4.6) | 8.9 (5.2)
  Day 21 | 4.40 (4.4) | 8.5 (6.2)
  Day 28 | 4.1 (4.7) | 8.0 (6.1)
Statistical Analysis 1: Comparison: Acupuncture vs Placebo Group; Test type: Superiority or Other; p = 0,05, ANOVA

3. Secondary Outcome: Quality of Life Assessed on the SF-36
Description: Questionnaire Short-form-36 is a widely used generic health status questionnaire, validated for Portuguese with eight components and each components with scores from 0 to 100: higher scores denote greater quality of life.
Time Frame: Days 0, 3, 7, 14, 21 and 28
Population: Intention to treat analysis (ITT)
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scale
Arm/Group | Acupuncture | Placebo Group
Number analyzed (Participants) | 40 | 40
Number analyzed (scale) | 40 | 40
scores on a scale
  Day 0 Functional Capacity | 46.4 (22.7) | 55.8 (19.2)
  Day 3 Functional Capacity | 58.5 (25.7) | 60.6 (19.6)
  Day 7 Functional Capacity | 68.8 (22.3) | 66.6 (17.1)
  Day 14 Functional Capacity | 78.6 (20.8) | 71.6 (20.8)
  Day 21 Functional Capacity | 81.8 (17.6) | 71.4 (21.7)
  Day 28 Functional Capacity | 84.0 (19.8) | 70.9 (22.5)
  Day 0 limitation in physical aspects | 18.1 (26.5) | 16.3 (26.3)
  Day 3 limitation in physical aspects | 35.6 (37.9) | 30.6 (33.2)
  Day 7 limitation in physical aspects | 53.1 (39.7) | 43.8 (40.7)
  Day 14 limitation in physical aspects | 70.6 (36.2) | 55.0 (35.0)
  Day 21 limitation in physical aspects | 75.6 (33.7) | 56.3 (39.9)
  Day 28 limitation in physical aspects | 78.8 (31.8) | 55.8 (38.3)
  Day 0 Pain | 27.6 (17.9) | 28.8 (19.1)
  Day 3 Pain | 46.1 (24.9) | 44.8 (19.4)
  Day 7 Pain | 54.8 (20.0) | 51.5 (21.4)
  Day 14 Pain | 64.9 (20.3) | 53.6 (19.2)
  Day 21 Pain | 69.3 (22.7) | 54.6 (24.7)
  Day 28 Pain | 67.8 (26.1) | 56.5 (23.4)
  Day 0 General Health State | 54.2 (25.7) | 56.5 (24.9)
  Day 3 General Health State | 60.5 (23.0) | 62.0 (22.4)
  Day 7 General Health State | 59.6 (25.9) | 63.7 (23.1)
  Day 14 General Health State | 66.6 (20.9) | 60.4 (23.3)
  Day 21 General Health State | 66.7 (22.2) | 58.4 (23.1)
  Day 28 General Health State | 69.0 (22.9) | 63.4 (22.6)
  Day 0 Vitality | 49.4 (25.3) | 47.6 (17.3)
  Day 3 Vitality | 56.4 (24.3) | 54.3 (20.0)
  Day 7 Vitality | 60.9 (23.1) | 57.1 (22.3)
  Day 14 Vitality | 69.3 (19.4) | 52.8 (24.1)
  Day 21 Vitality | 68.2 (20.4) | 56.3 (25.5)
  Day 28 Vitality | 69.6 (23.2) | 58.8 (24.0)
  Day 0 Social Aspects | 62.5 (34.6) | 65.9 (32.3)
  Day 3 Social Aspects | 76.9 (27.7) | 75.6 (29.7)
  Day 7 Social Aspects | 80.3 (27.9) | 80.9 (29.6)
  Day 14 Social Aspects | 89.4 (17.8) | 76.6 (31.9)
  Day 21 Social Aspects | 90.9 (17.0) | 79.4 (28.9)
  Day 28 Social Aspects | 89.7 (17.4) | 82.5 (25.9)
  Day 0 Emotional Aspects | 57.5 (41.3) | 62.5 (40.1)
  Day 3 Emotional Aspects | 73.3 (37.1) | 71.7 (40.3)
  Day 7 Emotional Aspects | 80.0 (33.6) | 78.3 (38.2)
  Day 14 Emotional Aspects | 84.2 (32.0) | 80.0 (30.9)
  Day 21 Emotional Aspects | 87.5 (24.7) | 73.3 (37.1)
  Day 28 Emotional Aspects | 81.7 (30.1) | 76.7 (36.4)
  Day 0 Mental Health | 54.3 (22.0) | 58.5 (19.7)
  Day 3 Mental Health | 63.1 (22.8) | 62.9 (21.3)
  Day 7 Mental Health | 67.4 (19.2) | 66.3 (21.0)
  Day 14 Mental Health | 68.5 (19.5) | 65.1 (21.3)
  Day 21 Mental Health | 69.3 (20.6) | 63.7 (25.2)
  Day 28 Mental Health | 66.4 (22.5) | 65.2 (22.8)

4. Secondary Outcome: Likert Improvement Assessment Scale
Description: Likert improvement assessment scale is based on the patient's opinion (LIKERT P) and assessor's opinion (LIKERT A), categorized in 1=MB (much better), 2=SB (slightly better), 3=NC (no change), 4=SW (slightly worse) and 5=MW (much worse). This scale was was applied to each day of assessment. The numbers in the category titles represent the different days.
Time Frame: Days 0, 3, 7, 14 and 21
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Acupuncture | Placebo Group
Number analyzed (Participants) | 40 | 40
scores on a scale
  Likert 0 P | 1.6 (0.54) | 2.15 (0.66)
  Likert 0 A | 1.6 (0.63) | 2.0 (0.78)
  Likert 3 P | 1.67 (0.72) | 2.27 (0.71)
  Likert 3 A | 1.62 (0.66) | 2.17 (0.81)
  Likert 7 P | 1.67 (0.72) | 2.20 (0.79)
  Likert 7 A | 1.55 (0.67) | 2.07 (0.91)
  Likert 14 P | 1.77 (0.73) | 2.05 (0.71)
  Likert 14 A | 1.65 (0.73) | 2.12 (0.82)
  Likert 21 P | 1.65 (0.8) | 2.07 (0.88)
  Likert 21 A | 1.62 (0.8) | 1.95 (0.81)

5. Secondary Outcome: Number of Anti-inflammatory Tablets Taken
Description: Number of 50 mg sodium diclofenac pills taken per day
Time Frame: Days 3,7,14,21 and 28
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: number of pills/day
Arm/Group | Acupuncture | Placebo Group
Number analyzed (Participants) | 40 | 40
number of pills/day
  Day 3 | 1.5 (2.6) | 2.6 (2.8)
  Day 7 | 1.9 (3.6) | 4.2 (4.7)
  Day 14 | 1.3 (3.1) | 3.3 (6.0)
  Day 21 | 1.2 (2.8) | 3.7 (5.2)
  Day 28 | 1.1 (2.7) | 2.3 (3.9)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected during de follow-up (28 days).
Description: 80 patients were evaluated in the end of the study and non-serious adverse events were observed.
Arm/Group | Acupuncture | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No